CLINICAL TRIAL: NCT01453413
Title: Blood Glucose Testing and You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CTD PRO 2011-003-01
Record Dates: First submitted 2011-09-30; First posted 2011-10-17 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- People with type 2 diabetes (Other): People with type 2 diabetes who were in attendance at a diabetes conference were asked for their perceived Blood Glucose (BG) value. Then, after staff measured BG on a Blood Glucose meter, subjects were informed of their BG value.
  Interventions: Other: Blood Glucose meter

INTERVENTIONS:
Other: Blood Glucose meter — Staff tested subject Blood Glucose using a Blood Glucose meter.
  Other Names: Contour® Blood Glucose Meter

SUMMARY:
The purpose of this study is to determine the difference between self-reported, estimated blood glucose level versus blood glucose levels measured with a Blood Glucose Meter.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 years of age and above
2. Type 2 diabetes
3. Able to speak, read, and understand English
4. Willing to complete all study procedures

Exclusion Criteria:

1. Type 1 diabetes
2. Currently a user of continuous glucose monitoring system
3. Currently pregnant
4. Hemophilia or any other bleeding disorder
5. Employee of competitive medical device company
6. Cognitive disorder or other condition which, in the opinion of the investigator (or designee), would put the person at risk or seriously compromise the integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Edelman, MD, Principal Investigator — Founder TCOYD
Locations (2):
- United States (2):
  - TCOYD at San Diego Convention Center, San Diego, California
  - TCOYD Conference at Tampa Convention Center, Tampa, Florida

REFERENCES:
- [Derived] Pettus J, Stenger P, Schachner HC, Dunne N, Parkes JL, Pardo S, Edelman SV. Testing versus guessing blood glucose values: impact on self-care behaviors in type 2 diabetes. Curr Med Res Opin. 2014 Sep;30(9):1795-802. doi: 10.1185/03007995.2014.929097. Epub 2014 Jun 30. PMID 24889281

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Type 2 Diabetes: Perceived BG value versus measured BG for people with type 2 diabetes who are in attendance at a diabetes conference
Period: Overall Study
Arm/Group | People With Type 2 Diabetes
Started | 297
Completed | 297
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- People With Type 2 Diabetes: People with type 2 diabetes who were in attendance at a diabetes conference were asked for their perceived Blood Glucose (BG) value. Then, after staff measured BG on Contour® Blood Glucose meter, subjects were informed of their BG value. Three subjects were excluded from all analyses due to inconsistencies in responses to inclusion / exclusion questions. So 294 subjects were included in demographics analyses.
Arm/Group | People With Type 2 Diabetes
Number analyzed (Participants) | 294
Age Continuous [Mean (Full Range); unit: years] | 59 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 117
Region of Enrollment [Number; unit: participants]
  United States | 294

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Outside Specified Blood Glucose (BG) Range -Estimated Versus Measured Blood Glucose
Description: The percent of subjects whose estimated blood glucose values are different than meter BG values. A calculation was performed to determine the percent of subjects whose estimated BG values are > +/-20% different than meter BG values when samples have BG >=75mg/dL or > +/- 15mg/dL different than meter BG values when samples have BG <75mg/dL, as measured by fingerstick CONTOUR®.
Time Frame: 1 visit 15-20 minutes
Population: Three subjects were excluded from analyses due to inconsistencies in responses to inclusion/exclusion questions(297-3=294). Eight subjects were excluded from BG analyses because they did not have both an estimated BG value and a meter result (294-8=286)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | People With Type 2 Diabetes
Number analyzed (Participants) | 286
percentage of subjects | 45.80 [40.12 to 51.60]

2. Secondary Outcome: Percent of Subjects Outside a Second Specified Blood Glucose (BG) Range -Estimated Versus Measured Blood Glucose
Description: The percent of subjects whose estimated blood glucose values are different than meter BG values. A calculation was performed to determine the percent of subjects whose estimated BG values are > +/-15% different than meter BG values when samples have BG >=100 mg/dL or > +/- 15 mg/dL different than meter BG values when samples have BG <100 mg/dL, as measured by fingerstick CONTOUR®.
Time Frame: 1 visit 15-20 minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | People With Type 2 Diabetes
Number analyzed (Participants) | 286
percentage of subjects | 57.69 [51.90 to 63.28]

ADVERSE EVENTS:
Arm/Group | People With Type 2 Diabetes
Serious Adverse Events (participants affected / at risk) | 0/297
Other Adverse Events (participants affected / at risk) | 3/297
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | People With Type 2 Diabetes (N=297)
hypoglycemia (Endocrine disorders) | 3 (3) — Non-serious, mild, anticipated, Not device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days